CLINICAL TRIAL: NCT01988792
Title: Human Milk Fortification and Feeding Intolerance in Very Low Birth Weight Neonates
Brief Title: Human Milk Fortification in Very Low Birth Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-02741-FB; 8671-2075 (Other Grant/Funding Number: Mead Johnson and Company LLC)
Record Dates: First submitted 2013-11-12; First posted 2013-11-20 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Premature; Infant; Enteral Nutrition; Human Milk; Fortification
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fortification at 20 ml/kg/day feeding volume (Active Comparator): Human milk fortifiers will be added to the human milk when neonates reach to feeding volume of 20 ml/kg/day.
  Interventions: Dietary Supplement: Human milk fortifiers
- Fortification at 100 ml/kg/day feeding volume (Active Comparator): human milk fortifiers will be added to the human milk when neonates reach to feeding volume of 100 ml/kg/day.
  Interventions: Dietary Supplement: Human milk fortifiers

INTERVENTIONS:
Dietary Supplement: Human milk fortifiers

SUMMARY:
The purpose of this study to find out how safely we can add extra nutrients to human milk at different feeding volume.

DETAILED DESCRIPTION:
Very low birth weight babies (weight less than three pounds and three ounces) are extremely fragile and lacking important nutrition due to premature birth. They need enough calories for catch-up growth. Giving adequate nutrition is very important for their growth and development. Human milk is the best food, however it is not enough to provide all the required calories and nutrients for catch up growth and maintain adequate strength of the bones (bone mineralization). For premature babies, extra nutrients (human milk fortifier) are usually added to the human milk to provide adequate nutrition. These extra nutrients will be derived from cow's milk. Currently, a practice of fortifying human milk varies. There is no clear information when to start adding extra nutrients to human milk.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants who receive human milk (mother's milk or banked donor human milk).

Exclusion Criteria:

* Major congenital anomalies such as cardiac defect, neural tube defect, chromosomal abnormality and gastrointestinal defect.
* Died or extended to die within 48 hours of life

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The days to reach full enteral feeding volume (140 ml/kg/day). | 4 - 6 weeks

SECONDARY OUTCOMES:
Neonatal Outcomes | until 36 weeks PMA
  Necrotizing Enterocolitis
Neonatal Outcomes | until 36 weeks PMA
  Chronic Lung Disease
Neonatal Outcomes | Until full feeding volume
  Feeding intolerance
Neonatal Outcomes | Until full feeding volume
  Parental nutrition days
Neonatal Outcomes | until 36 weeks PMA
  Ventilator days
Neonatal Outcomes | until 4 weeks of life
  Protein and caloric intake
Neonatal Outcomes | until 4 weeks of life
  Growth anthropometry

CONTACTS AND LOCATIONS:
Overall Officials: Sanket D Shah, MBBS, Principal Investigator — UTHSC, Memphis, TN; Ajay J Talati, MD, Principal Investigator — UTHSC, Memphis, TN
Locations (1):
- University of Tennessee, Health Science Center, The Regional Medical Center, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Shah SD, Dereddy N, Jones TL, Dhanireddy R, Talati AJ. Early versus Delayed Human Milk Fortification in Very Low Birth Weight Infants-A Randomized Controlled Trial. J Pediatr. 2016 Jul;174:126-131.e1. doi: 10.1016/j.jpeds.2016.03.056. Epub 2016 Apr 23. PMID 27112041